CLINICAL TRIAL: NCT04641845
Title: The Effects of Small Variations in Shoe Heel Height on Gait in People With a Transtibial Amputation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 638_Heel Height Amputation
Record Dates: First submitted 2020-11-04; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Lower Limb Amputation Below Knee (Injury)
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Experimental repeated measures study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heel height increases (Experimental): All participants consecutively walked with four heel height conditions (0 millimeter, 3 millimeter, 5 millimeter and 8 millimeter). The order of the heel height conditions was randomized.
  Interventions: Other: Cork inlay wedge

INTERVENTIONS:
Other: Cork inlay wedge

SUMMARY:
Prosthetic alignment is important for walking function and walking comfort in people with a transtibial amputation (TTA). Prosthetic alignment is defined as the position of prosthetic parts relative to the body and to each other. A suboptimal alignment decreases stability and increases energy use during walking. Therefore, finding the optimal alignment is an important aspect of rehabilitation. Shoe heel height is considered to influence prosthetic alignment, walking comfort and gait symmetry in people with a TTA. Unfortunately, research on the effect of heel height is scarce and no evidence is available on the effects of variations smaller than 20 mm. However, these small heel height variations between store-bought shoes are often overlooked by people with an amputation and may cause secondary musculoskeletal problems in the long term. To increase the knowledge on this topic, this study aims to examine the effects of small increases in heel height on gait symmetry in people with a TTA and healthy individuals. It was expected that higher heel height would cause more asymmetry in gait and lower walking comfort. People with a TTA were expected to be affected more by heel height changes than healthy individuals.

DETAILED DESCRIPTION:
Optimal prosthetic alignment is essential to achieve a functional gait pattern in people with a transtibial amputation (TTA). A suboptimal alignment decreases stability, increases the metabolic costs of walking, and increases the risk of secondary musculoskeletal and stump problems. Prosthetic alignment is defined as the position of the prosthetic parts relative to the body and to each other. Dynamic alignment of the prosthesis, especially the 'fine tuning' of the prosthesis based on the patient's needs, is a continuous process during rehabilitation.

Throughout the entire alignment process the prosthetists takes the shoe heel height of the patient into account. Moreover, patients are advised to search for a similar heel height when purchasing new shoes. However, prosthetic walkers frequently report complaints during their follow-up visits with their prosthetist or rehabilitation physician that possibly are related to prosthetic misalignment. Although several studies describe the effects of heel height on gait in healthy individuals, our knowledge about the effects of heel height within the TTA population is still limited to one study examining heel height changes of 20 millimeter. The variation in heel height of commercially available shoes is often smaller, and therefore easily overlooked by people with a TTA. Since it is not clear what the effects of smaller heel height variations on the gait pattern are, additional research is needed to enable prosthetists and therapists to better advise their patients.

Therefore, the primary objective was to examine the effect of small increases in heel height on gait symmetry in people with a TTA. It was expected that a larger increase in heel height would result in more gait asymmetry and lower walking comfort. In addition, healthy individuals were included in whom smaller effects of the heel height changes were expected.

ELIGIBILITY:
Inclusion Criteria:

* had their prosthesis for at least one year (participants with a TTA)

Exclusion Criteria:

* (other) neurological or orthopaedic impairments affecting walking ability
* surgery on the lower extremities within the last six months
* the use of a walking aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Symmetry of the centre of pressure velocity (VCOP symmetry) | On average, during 10 minutes.
  Symmetry of the VCOP trajectories during the stance phase of gait between the prosthetic leg and sound leg (participants with TTA), or the right and left leg (healthy individuals), calculated with the root mean square.

SECONDARY OUTCOMES:
Step length symmetry | On average, during 10 minutes
  Ratio index of step length between left and right leg.
Single leg stance time symmetry | On average, during 10 minutes
  Ratio index of single leg stance time between left and right leg.
Double limb support symmetry | On average, during 10 minutes
  Ratio index of percentage of double limb support between left and right leg (Xright/(Xright+Xleft).
Experienced walking comfort | On average, at 2.5 minutes, 5 minutes, 7.5 minutes and 10 minutes.
  Experienced walking comfort is measured with a visual analog scale (VAS) of 10 centimeters (lowest score is 0, highest score is 10).

CONTACTS AND LOCATIONS:
Overall Officials: Noël LW Keijsers, PhD, Study Chair — Sint Maartenskliniek

IPD SHARING:
Plan to Share IPD: No